CLINICAL TRIAL: NCT05588531
Title: Study on Tolerance, Pharmacokinetics and Drug Interaction of YK-1169 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: NJLBW-YK-1169
Record Dates: First submitted 2022-08-19; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Pharmacokinetics
Keywords: YK-1169
MeSH Terms: interventions — Injections; avibactam

STUDY DESIGN:
Intervention Model Description: The whole trial is conducted by dose escalation from low to high.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- YK-1169 0.5g (containing cefepime 0.4g, avibactam 0.1g) (Active Comparator): Four healthy subjects in group A1, two males and two females, without control, were administered the test drug
  Interventions: Drug: Group 1:YK-1169
- YK-1169 1.25 g (containing cefepime 1.0 g and avibactam 0.25 g) (Active Comparator): 12 healthy subjects, of whom 10 subjects were administered the investigational product and 2 subjects were administered placebo, half males and half females
  Interventions: Drug: Group 2:YK-1169/Placebo Injection
- YK-1169 2.5g (containing cefepime 2.0g and avibactam 0.5g) (Active Comparator): 12 healthy subjects, of whom 10 subjects were administered the investigational product and 2 subjects were administered placebo, half males and half females
  Interventions: Drug: Group 3:YK-1169/Placebo
- YK-1169 3.75g (containing cefepime 3.0g and avibactam 0.75g) (Placebo Comparator): 12 healthy subjects, of whom 10 subjects were administered the investigational product and 2 subjects were administered placebo, half males and half females
  Interventions: Drug: Group 4:YK-1169/Placebo
- YK-1169 5.0g (containing cefepime 4.0g and avibactam 1.0g) (Active Comparator): 8 healthy subjects, 6 of whom were administered the investigational product and 2 of whom were administered placebo, half males and half females
  Interventions: Drug: Group 5:YK-1169/Placebo Injection
- Drug Interaction Studies (Active Comparator): 18 subjects (single gender not less than 1/3) were randomly divided into D1, D2 and D3 groups, 6 subjects for each group
  Interventions: Drug: Group 1:YK-1169; Drug: Group 6:YK-1169/Cefepime hydrochloride for injection/Avibactam for injection

INTERVENTIONS:
Drug: Group 1:YK-1169 — YK-1169 0.5g (containing cefepime 0.4g, avibactam 0.1g) single intravenous infusion for 2 hours
  Arms: Drug Interaction Studies; YK-1169 0.5g (containing cefepime 0.4g, avibactam 0.1g)
Drug: Group 2:YK-1169/Placebo Injection — YK-1169 1.25g (containing cefepime 1.0g, avibactam 0.25g) / placebo single intravenous infusion for 2 hours
  Arms: YK-1169 1.25 g (containing cefepime 1.0 g and avibactam 0.25 g)
Drug: Group 3:YK-1169/Placebo — On the first day, YK-1169 2.5 g (containing cefepime 2.0 g, avibactam 0.5g) was single intravenously infused for 2 h. On the third day, YK-1169 2.5 g (containing cefepime 2.0 g, avibactam 0.5g) was single intravenous infusion for 2 h, three times a day at 8-h intervals, until the morning dose on the tenth day
  Arms: YK-1169 2.5g (containing cefepime 2.0g and avibactam 0.5g)
Drug: Group 4:YK-1169/Placebo — On the first day, YK-1169 3.75 g (containing cefepime 3.0 g, avibactam 0.75g) was single intravenously infused for 2 h. On the third day, YK-1169 3.75 g (containing cefepime 3.0 g, avibactam 0.75g) was single intravenous infusion for 2 h, three times a day at 8-h intervals, until the morning dose on the tenth day
  Arms: YK-1169 3.75g (containing cefepime 3.0g and avibactam 0.75g)
Drug: Group 5:YK-1169/Placebo Injection — YK-1169 5.0g (containing cefepime 4.0g, avibactam 1.0g) / placebo single intravenous infusion for 2 hours
  Arms: YK-1169 5.0g (containing cefepime 4.0g and avibactam 1.0g)
Drug: Group 6:YK-1169/Cefepime hydrochloride for injection/Avibactam for injection — YK-1169 2.5g (containing cefepime 2.0g, avibactam 0.5g)/cefepime hydrochloride for injection 2.0g/avibactam for injection 0.5g, three-cycle three-cross single intravenous infusion for 2 hours
  Arms: Drug Interaction Studies

SUMMARY:
To evaluate the safety and tolerability of multiple doses of YK-1169 in healthy subjects, the pharmacokinetic characteristics of multiple doses in healthy subjects, and the drug interaction between cefepime and avibactam.

DETAILED DESCRIPTION:
A randomized, single-blind, placebo-controlled, dose-escalation, single-center clinical trial design was used. A total of 5 dose groups A1, A2, A3, A4 and A5 were set in the test, including A1 YK-1169 0.5g group (containing cefepime 0.4g and avibactam 0.1g), A2 YK-1169 1.25g group (containing cefepime 1.0g and avibactam 0.25g), A3 YK-1169 2.5g (containing cefepime 2.0g and avibactam 0.5g), A4 YK-1169 3.75g (containing cefepime 3.0g and avibactam 0.75g) and A5 YK-1169 5.0g (containing cefepime 4.0g and avibactam 1.0g).

A single-center, randomized, open, three-period three-crossover 3 × 3 Latin square trial design was used. To study the effect of intravenous infusion of this product, cefepime for injection or avibactam for injection on the disposition process of the drug in the human body, so as to study whether there is a pharmacokinetic drug interaction in this product.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects aged 18 to 45 years (including the cut-off value), both men and women;
2. body mass index (BMI) 19.0-28.0 kg/m2 (including the cut-off value);
3. fully understand the purpose of the trial, basically understand the pharmacological effects of the investigational drug and possible risks, voluntarily sign the informed consent form;
4. be able to communicate well with the investigator, and understand and abide by the requirements of this study.

Exclusion Criteria:

1. participate in any drug clinical trials or use of study drugs within 3 months before the use of study drugs;
2. have a history of respiratory system, digestive system, cardiovascular system, endocrine system, urinary system, nervous system (such as epilepsy, etc.), hematology, immunology (including personal or family history of hereditary immunodeficiency), metabolic abnormalities and the investigator believes that there is still clinical significance;
3. allergic to penicillins, allergic to cephalosporins, allergic to amoxicillin clavulanate potassium tablets or their excipients, or a history of drug, food or other substance allergy;
4. can not tolerate intravenous puncture or have a history of halo, fainting needle;
5. received surgery within 6 months before the use of study drugs that will affect drug distribution, metabolism, excretion; or received surgery within 4 weeks before the use of study drugs; or plan to undergo surgery during the study period; -
6. Use of any drugs (including Chinese herbal medicine, health products, etc.) within 14 days before the use of the study drug;
7. Vaccination or live attenuated vaccine within 14 days before the use of the study drug, or plan to vaccinate during the trial;
8. Blood donation or massive blood loss (> 400 mL) within 3 months before the use of the study drug, receiving blood transfusion or use of blood products, or intend to donate blood or blood components during the trial or within 3 months after the end of the trial;
9. Drug abusers or use of soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the use of the study drug;
10. Smokers or smokers who smoke more than 5 cigarettes per day for 3 months before the use of the study drug, or can not stop using any tobacco products during the trial;
11. habitual drinking, tea, coffee and/or caffeine-containing beverages and do not agree to stop eating the above diet during the trial;
12. special requirements for diet, can not comply with the unified diet, or lactose intolerance;
13. volunteers (or their partners) during the trial to 3 months after the end of the trial have a pregnancy plan, sperm donation and egg donation plan, or reluctant to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, contraceptive rings, partner ligation, etc.);
14. female volunteers are pregnant or lactating women; or have non-protective sex within 2 weeks before the use of the study drug; or use oral contraceptives within 30 days before the use of the study drug or use of long-acting estrogen or progestogen injection or implants within 6 months before the use of the study drug; 15. physical examination, 12-lead electrocardiogram, vital signs, abdominal ultrasound, chest X-ray, laboratory tests are abnormal clinical significance (subject to the clinician 's judgment);

16. Volunteers may not be able to complete this study for other reasons or have other reasons for not being suitable for the trial judged by the investigator; 17. First cycle admission examination vital signs abnormal clinical significance, drug screening positive, alcohol test positive or female pregnancy test abnormal clinical significance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
According to Common Terminology Criteria for Adverse Events Version 5.0, the incidence and frequency of AEs and SAEs will be statistically analyzed | Through study completion, an average of 1 month.
  Descriptive analysis was used to calculate the incidence of adverse events and adverse reactions, and the number and frequency of occurrence of various adverse events and adverse reactions.
clinical adverse events | Through study completion, an average of 1 month.
  Descriptive analysis was used to analyze the relationship and outcome between the degree and duration of adverse events and the drug on a case-by-case basis
body temperature (frontal temperature) | Through study completion, an average of 1 month.
  Abnormal body temperature (frontal temperature) and body temperature (℃) before and after administration will be analyzed on a case-by-case basis
Pulse | Through study completion, an average of 1 month.
  Abnormal pulse before and after dosing will be analyzed on a case-by-case basis. Pulse (beats/min)
sitting blood pressure | Through study completion, an average of 1 month.
  Abnormal blood pressure before and after dosing will be analyzed on a case-by-case basis. Blood pressure (MmHg)
physical examination | Through study completion, an average of 1 month.
  Abnormalities before and after administration of physical examination were analyzed on a case-by-case basis
laboratory tests | Through study completion, an average of 1 month.
  Abnormalities before and after administration in laboratory tests were analyzed on a case-by-case basis
12-lead ECG | Through study completion, an average of 1 month.
  Abnormalities before and after 12-lead ECG administration were analyzed on a case-by-case basis
premature withdrawal | Through study completion, an average of 1 month.
  Analysis of early withdrawals on a case-by-case basis

SECONDARY OUTCOMES:
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: Cmax | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: Cmax
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: Tmax | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: Tmax
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: AUC | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: AUC
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: t1/2 | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: t1/2
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: CL | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: CL
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: VZ | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: VZ
The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: λz | Single dose: within 1 hour before to 24 hours after dosing on Day 1.Drug Interactions: Within 1 hour prior to dosing on Day 1 through 24 hours postdose of each cycle
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. The main pharmacokinetic parameters evaluated in the single-dose and drug-drug interaction studies included: λz
Cumulative urinary excretion ratio, etc. in 2.5 g single dose group of YK-1169 | Single dose: within 1 hour before to 24 hours after dosing on Day 1
  Pharmacokinetic parameters were calculated using WinNonlin 8.2 (or higher) software from Certara, USA. Calculated cumulative urinary excretion ratio, etc. for 2.5 g single dose of YK-1169
Main pharmacokinetic parameters evaluated in multiple dose studies included: C min, ss | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included: C min, ss
Main pharmacokinetic parameters evaluated in multiple dose studies included: C max,ss | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included: C max,ss
Main pharmacokinetic parameters evaluated in multiple dose studies included: Tmax,ss | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included: Tmax,ss
Main pharmacokinetic parameters evaluated in multiple dose studies included:AUC | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included:AUC
Main pharmacokinetic parameters evaluated in multiple dose studies included:Cav,ss | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included:Cav,ss
Main pharmacokinetic parameters evaluated in multiple dose studies included:t1/2 | Multiple dose: within 1 hour before dosing on Day 1 to D9 (24 hours after dosing on D8).
  Main pharmacokinetic parameters evaluated in multiple dose studies included:t1/2

CONTACTS AND LOCATIONS:
Locations (1):
- 辛玉霞, Nanjing, Jiangsu, China